CLINICAL TRIAL: NCT01642602
Title: A Phase 2 Open-Label, Multicenter, 4-Week Study to Assess the Safety and Effectiveness of Daily Oral Administration of Dexlansoprazole Delayed-Release Capsules for Relief of Heartburn, in Adolescent Subjects Aged 12 to 17 Years With Symptomatic Non-Erosive Gastroesophageal Reflux Disease
Brief Title: Safety and Efficacy of Dexlansoprazole Delayed-Release Capsules in Treating Symptomatic Non-Erosive Gastroesophageal Reflux Disease in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-390MR_206; U1111-1128-5977 (Registry Identifier: WHO); 2012-001680-72 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg delayed-release capsules orally once daily for up to 4 weeks.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release capsules.
  Other Names: Dexilant; TAK-390MR

SUMMARY:
The purpose of this study was to assess the safety and effectiveness of once daily oral administration of dexlansoprazole delayed-release capsules in adolescent participants with symptomatic non-erosive gastroesophageal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant and parent(s) or legal guardian are capable of understanding and complying with protocol requirements.
2. Prior to any study-specific procedures being performed, the informed consent and the assent form, according to local country requirements, must be signed and dated by parent(s) or legal guardian and by the participant, respectively.
3. The participant has a medical history of symptoms of GERD for at least 3 months prior to Screening (signed informed consent and assent if applicable), as assessed by the investigator.
4. The participant has met the electronic diary qualification criteria as assessed by the electronic daily diary defined as follows: heartburn (burning or hurting in your throat, chest, or stomach) on at least 3 of 7 days.
5. The participant has non-erosive GERD with no evidence of definite endoscopic esophageal mucosal breaks as described in the Los Angeles Classification of Esophagitis at the screening endoscopy
6. The participant is male or female and aged 12 to 17 years, inclusive.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent and assent throughout the duration of the study and for 30 days after last dose of study medication.
8. A female participant of childbearing potential who is or may become sexually active agrees to routinely use adequate contraception from the time of signing the informed consent and assent until 30 days after the last dose of study medication.

Exclusion Criteria:

1. Participant has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, or metabolic, endocrine or gastrointestinal disease, or serious allergy, asthma, or allergic skin rash that suggests clinically significant, uncontrolled underlying disease or condition (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. The participant has a co-existing disease affecting the esophagus), (eg, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
3. The participant has a known history of Barrett's with dysplastic changes in the esophagus.
4. The participant has a known history of eosinophilic esophagitis (EoE) or endoscopic findings suggestive of EoE.
5. The participant has a history of celiac disease or the participant tests positive for tTG antibody.
6. The participant has active gastric or duodenal ulcers within 4 weeks prior to Day -1.
7. Participant has any finding in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
8. Participant has taken any PPI within 1 week (7 days) prior to the Screening Visit.
9. The participant has a history of hypersensitivity or allergies to dexlansoprazole or any component of dexlansoprazole or any PPI (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole or antacid containing Mg(OH)2 and / or Al (OH)3 or simethicone.
10. The participant is required to take excluded medications or it is anticipated that the participant will require treatment with at least one of the disallowed concomitant medications during the study evaluation period as specified in the Excluded Medications and Treatments Section 7.3.
11. The participant has a history of malignant disease (except basal cell carcinoma) within 5 years prior to Screening.
12. The participant has a condition that may require inpatient surgery during the course of the study.
13. The participant requires dilatation of esophageal strictures and/or strictures preventing passage of the endoscope during the Screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
14. The participant is known to be positive for human immunodeficiency virus (HIV).
15. The participant has current or clinical history of Zollinger-Ellison syndrome or other hypersecretory condition.
16. The participant has a history of gastric, duodenal or esophageal surgery except simple oversew of an ulcer. A history of gastric tube and/or percutaneous endoscopic gastrostomy (PEG) placement is allowed.
17. The participant had an acute upper gastrointestinal hemorrhage within 4 weeks prior to endoscopy.
18. The participant has donated or lost ≥300 mL blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
19. The participant has a known history of alcohol abuse or illegal drug use within the past 12 months prior to the first dose of study drug.
20. The participant has any Screening Visit 1 abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (×ULN), or total bilirubin >2.0 mg/dL with AST/ALT elevated above the limits of normal values.
21. If female, the participant is pregnant or lactating or intending to become pregnant before, during or within 30 days after last dose of study medication; or intending to donate ova during such time period.
22. If male, the participant intends to donate sperm during the course of this study or within 30 days after last dose of study drug.
23. The participant, participant's Parent(s) or Legal Guardian is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent and assent under duress. Students of the institution/research facility who are under the supervision of, or in a subordinate role to, the investigator are also ineligible.
24. The participant or participant's Parent(s) or Legal Guardian, in the opinion of the investigator, is unlikely to comply with the protocol requirements or is unsuitable for any other reason.
25. The participant has participated in another clinical study and/or has received any investigational compound within 30 days prior to Screening.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research and Development Center, Inc.
Locations (64):
- United States (35):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Los Angeles, California
  - San Francsco, California
  - Centennial, Colorado
  - Thornton, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Flint, Michigan
  - Plymouth, Minnesota
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Mays Landing, New Jersey
  - Brooklyn, New York
  - Huntsville, North Carolina
  - Toledo, Ohio
  - Youngstown, Ohio
  - Greenville, South Carolina
  - Kingsport, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Norfolk, Virginia
- Brussels, Belgium
- Brazil (4):
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
- Hungary (6):
  - Debrecen
  - Győr
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Veszprém
- Italy (3):
  - Bari, Bari
  - Messina, Messina
  - Roma, Roma
- Mexico (3):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
- Poland (7):
  - Bydgoszcz
  - Krakow
  - Rzeszów
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
- Portugal (5):
  - Amadora
  - Braga
  - Coimbra
  - Lisbon
  - Porto

REFERENCES:
- [Derived] Gold BD, Pilmer B, Kierkus J, Hunt B, Perez MC, Gremse D. Dexlansoprazole for Heartburn Relief in Adolescents with Symptomatic, Nonerosive Gastro-esophageal Reflux Disease. Dig Dis Sci. 2017 Nov;62(11):3059-3068. doi: 10.1007/s10620-017-4743-3. Epub 2017 Sep 15. PMID 28916953
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 36 sites in the United States, Belgium, Hungary, Italy, Poland, Portugal, Brazil, and Mexico from 22 June 2012 to 21 January 2014.
Pre-assignment Details: Adolescent participants (male or female), aged 12 to 17 years (inclusive) with symptomatic non-erosive gastrointestinal reflux disease were enrolled in 1 group and received dexlansoprazole 30 mg orally once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Dexlansoprazole 30 mg
Started | 104
Completed | 102
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set: All participants who received at least 1 dose of study drug and had post-baseline data (and baseline data if applicable) for the appropriate efficacy variable.
Arm/Group | Dexlansoprazole 30 mg
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.50)
Age, Customized [Number; unit: participants]
  12 to 14 years | 34
  15 to 17 years | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6
  White | 95
  Multiracial | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 19
  Non-Hispanic and Latino | 47
  Not Collected | 38
Weight [Mean (Standard Deviation); unit: kg] | 61.60 (14.393)
Height [Mean (Standard Deviation); unit: cm] | 163.1 (7.58)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.02 (4.434)
Smoking Classification [Number; unit: participants]
  Never Smoked | 103
  Ex-smoker | 1
H pylori Status [Number; unit: participants]
  Positive | 14
  Negative | 90

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Experience Each Treatment Emergent Adverse Event Experienced by ≥5% of Participants While Receiving Dexlansoprazole During the 4 Week Treatment Period
Description: A Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event (AE) that started or worsened on or after Study Day 1 (defined as first dose day), and no more than 30 days after the last dose of study drug.
Time Frame: 4 weeks
Population: Safety analysis set: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Dexlansoprazole 30 mg
Number analyzed (Participants) | 104
Percentage of participants
  Diarrhoea | 6.7
  Headache | 6.7

2. Secondary Outcome: The Percentage of Days With Neither Daytime Nor Nighttime Heartburn Over the 4 Weeks of Treatment
Description: Participants documented the presence or absence and the degree to which daytime and nighttime heartburn symptoms hurt daily in an electronic daily diary.
Time Frame: 4 weeks
Population: Full analysis set: All participants who received at least 1 dose of study drug and had post-baseline data (and baseline data if applicable) for the efficacy variable.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Dexlansoprazole 30 mg
Number analyzed (Participants) | 104
Percentage of days | 47.3 (32.18) [0 to 100]

ADVERSE EVENTS:
Time Frame: A Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event (AE) that started or worsened on or after Study Day 1 (defined as first dose day), and no more than 30 days after the last dose of study drug
Description: At each visit, the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole 30 mg
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 14/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 30 mg (N=104)
Diarrhoea (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.